CLINICAL TRIAL: NCT06397768
Title: Phase III, Randomized, Single-blind, Placebo-controlled, Multi-center Study to Evaluate Non-interference of Concomitant Administration of Routine Pediatric Vaccines on the Antibody Response of an Investigational Live-attenuated Respiratory Syncytial Virus (RSV) Vaccine in Healthy Infants and Toddlers (CORAL)
Brief Title: Co-administration Study of an Investigational Live-Attenuated Respiratory Syncytial Virus Vaccine in Infants and Toddlers
Acronym: CORAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAD00016; VAD00016 (Other: Sanofi Identifier); U1111-1290-7356 (Registry Identifier: ICTRP); 2024-000262-15 (EudraCT Number)
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: RSV Immunization
MeSH Terms: interventions — YM 534; Tetanus Toxoid; Hepatitis B Vaccines; Vaxelis; Poliovirus Vaccines; pentacel; Recombivax HB; Pneumococcal Vaccines; Rotavirus Vaccines; RotaTeq; Measles-Mumps-Rubella Vaccine; Herpes Zoster Vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * Blinding for vaccine group assignment: participants, parents or legally acceptable representatives (LAR) and laboratory personnel at the Sponsor
  * No blinding for study staff who prepare and administer the study interventions, investigators or Sponsor study staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Group 1- (RSVt vaccine concomitantly at 6 months) (Experimental): Participants will be administered RSVt vaccine concomitantly with routine pediatric vaccines, 2 doses, at age 6 months. Vaccines administered at age 6 months: RSVt Vaxelis or Pentacel and Recombivax HB, Prevnar 20, and RotaTeq. Placebo will be administered non-concomitantly at 7 months of age
  Interventions: Biological: RSVt vaccine; Biological: Diphtheria, tetanus, pertussis, poliomyelitis , Haemophilus influenzae type b, and hepatitis B vaccine; Biological: Diphtheria, tetanus, pertussis, Haemophilus influenzae type b and poliomyelitis vaccine; Biological: Hepatitis B vaccine; Biological: Streptococcus pneumoniae vaccine; Biological: Rotavirus vaccine; Biological: Placebo
- Cohort 1: Group 2- (RSVt vaccine non-concomitantly at 7 months) (Experimental): Participants will be administered RSVt vaccine non-concomitantly with routine pediatric vaccines, 2 doses, at age 7 months. Vaccines administered at age 6 months: Vaxelis or Pentacel and Recombivax HB, Prevnar 20, and RotaTeq. Placebo will be administered concomitantly at 6 months of age
  Interventions: Biological: RSVt vaccine; Biological: Diphtheria, tetanus, pertussis, poliomyelitis , Haemophilus influenzae type b, and hepatitis B vaccine; Biological: Diphtheria, tetanus, pertussis, Haemophilus influenzae type b and poliomyelitis vaccine; Biological: Hepatitis B vaccine; Biological: Streptococcus pneumoniae vaccine; Biological: Rotavirus vaccine; Biological: Placebo
- Cohort 2: Group 3- (RSVt vaccine concomitantly at 12 months) (Experimental): Participants will be administered RSVt vaccine concomitantly with routine pediatric vaccines, 2 doses, at age 12 months. Vaccines administered at age 6 months: M-M-R II, VARIVAX, and Prevnar 20. Placebo will be administered non-concomitantly at 13 months of age
  Interventions: Biological: RSVt vaccine; Biological: Streptococcus pneumoniae vaccine; Biological: Measles, mumps, and rubella vaccine; Biological: Varicella virus vaccine; Biological: Placebo
- Cohort 2: Group 4- (RSVt vaccine non-concomitantly at 13 months) (Experimental): Participants will be administered RSVt vaccine non-concomitantly with routine pediatric vaccines, 2 doses, at age 13 months. Vaccines administered at age 6 months: M-M-R II, VARIVAX, and Prevnar 20. Placebo will be administered concomitantly at 12 months of age
  Interventions: Biological: RSVt vaccine; Biological: Streptococcus pneumoniae vaccine; Biological: Measles, mumps, and rubella vaccine; Biological: Varicella virus vaccine; Biological: Placebo

INTERVENTIONS:
Biological: RSVt vaccine — Pharmaceutical form:Liquid for nasal spray-Route of administration:Intranasal
  Other Names: 534
Biological: Diphtheria, tetanus, pertussis, poliomyelitis , Haemophilus influenzae type b, and hepatitis B vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Vaxelis®
  Arms: Cohort 1: Group 1- (RSVt vaccine concomitantly at 6 months); Cohort 1: Group 2- (RSVt vaccine non-concomitantly at 7 months)
Biological: Diphtheria, tetanus, pertussis, Haemophilus influenzae type b and poliomyelitis vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Pentacel®
  Arms: Cohort 1: Group 1- (RSVt vaccine concomitantly at 6 months); Cohort 1: Group 2- (RSVt vaccine non-concomitantly at 7 months)
Biological: Hepatitis B vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: RECOMBIVAX HB® or alternate monovalent hepatitis B vaccine
  Arms: Cohort 1: Group 1- (RSVt vaccine concomitantly at 6 months); Cohort 1: Group 2- (RSVt vaccine non-concomitantly at 7 months)
Biological: Streptococcus pneumoniae vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: PREVNAR 20®
Biological: Rotavirus vaccine — Pharmaceutical form:Oral solution-Route of administration:Oral
  Other Names: RotaTeq®
  Arms: Cohort 1: Group 1- (RSVt vaccine concomitantly at 6 months); Cohort 1: Group 2- (RSVt vaccine non-concomitantly at 7 months)
Biological: Measles, mumps, and rubella vaccine — Pharmaceutical form:Lyophilized live virus for reconstitution -Route of administration:Subcutaneous or Intramuscular
  Other Names: M-M-R® II
  Arms: Cohort 2: Group 3- (RSVt vaccine concomitantly at 12 months); Cohort 2: Group 4- (RSVt vaccine non-concomitantly at 13 months)
Biological: Varicella virus vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Subcutaneous or Intramuscular
  Other Names: VARIVAX®
  Arms: Cohort 2: Group 3- (RSVt vaccine concomitantly at 12 months); Cohort 2: Group 4- (RSVt vaccine non-concomitantly at 13 months)
Biological: Placebo — Pharmaceutical form:Liquid for nasal spray-Route of administration:Intranasal

SUMMARY:
This study is a Phase III, randomized, single-blind, placebo-controlled, multi-center study to be conducted in healthy infants and toddlers which will be enrolled at approximately 6 months of age (Cohort 1) and approximately 12 months of age (Cohort 2). The primary objective of the study will be to assess non-inferiority of the RSV infant and toddler (RSVt) vaccine antibody response when administered concomitantly with routine pediatric vaccines at 6 months of age (Diphtheria and Tetanus Toxoids and Acellular Pertussis, Inactivated Poliovirus, Haemophilus b Conjugate and Hepatitis B Vaccine [Vaxelis® or Pentacel® and Recombivax HB®] Prevnar 20®, and RotaTeq®), and 12 months of age (M-M-R II, VARIVAX, and Prevnar 20 or per local country recommendations) compared to when administered non-concomitantly.

DETAILED DESCRIPTION:
The study duration is approximately 9 months for each participant.

* Cohort 1: Visits at 6, 7, and 8 and 9 months of age for both groups with visit at 10 months of age for Group 2 only
* Cohort 2: Visits at 12, 13, 14 and 15 months of age for both groups with visit at 16 months of age for Group 4 only
* Routine pediatric vaccines (authorized auxiliary medicinal products (AxMP) will be administered at 6 months in Cohort 1 and 12 months of age in Cohort 2, as per Advisory Committee on Immunization Practice (ACIP) or local country recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months for Cohort 1 and 12 months for Cohort 2 on the day of inclusion ("6 months" means from the day of the 6-month birthday to the day before the 7-month birthday and "12 months" means from the day of the 12-month birthday to the day before the 13-month birthday)
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* For Cohort 1: Infant received doses of vaccines containing hepatitis B, diphtheria, tetanus, pertussis, Haemophilus influenzae type B (Hib), and inactivated poliovirus vaccine (IPV) antigens, with Advisory Committee on Immunization Practice (ACIP) recommended vaccines. The last dose(s) of these vaccines must be at least 28 days before the first study visit
* Infant received the recommended doses of a recommended pneumococcal conjugate vaccine (as per local schedule) at least 28 days before the first study visit.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known previous infection with diphtheria, tetanus, Hib, measles, mumps, rubella, rotavirus, pneumococcus, polio, hepatitis B virus
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* History of medically diagnosed wheezing
* Any acute febrile illness in the past 48 hours that according to investigator judgment is significant enough to interfere with successful inoculation on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Probable or confirmed ongoing case of viral respiratory infection (including COVID 19, influenza, rhinovirus, etc.) at the time of enrollment. A prospective participant should not be included in the study until the respiratory infection has resolved.
* Member of a household that contains an immunocompromised individual, including, but not limited to:
* A person living with human immunodeficiency virus (HIV)
* A person who has received chemotherapy within the 12 months prior to study enrollment
* A person who has received (within the past 6 months) or is receiving (at the time of enrollment) immunosuppressant agents
* A person living with a solid organ or bone marrow transplant
* Potential close contact with other immunocompromised individual within 30 days after each vaccination as per investigator's discretion
* History of definitive contraindications to any of the concomitant vaccines that will be administered as part of the study protocol
* Participant's biological mother with previous receipt or planned administration of an investigational RSV vaccine during pregnancy and/or breastfeeding
* Receipt of any vaccine in the 4 weeks preceding RSVt vaccine administration or planned receipt of any vaccine outside of study protocol in the 4 weeks following RSVt vaccine administration, except for influenza and/or COVID-19 vaccination, which may be received at least 1 week before or 1 week after RSVt vaccine administration
* Previous receipt of an investigational RSV vaccine or receiving any anti RSV product (such as ribavirin or RSV immune globulin) at the time of enrollment
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of intranasal and intra-ocular medications within 3 days prior to study enrollment
* Previous receipt of an RSV monoclonal antibody within 6 months prior to the first study vaccine administration or planned receipt for duration of the study
* For Cohort 1: Prior receipt of routine 6-month pediatric vaccine doses (as per local schedule)
* For Cohort 2: Prior receipt of routine 12-month pediatric vaccine doses (as per local schedule)
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2226 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
RSV A serum neutralizing antibody titers at 28 days post dose 2 (D85) Groups 1 and 3 | Day 85
  Antibody titers at Day 85
RSV B serum neutralizing antibody titers at 28 days post dose 2 (D85) Groups 1 and 3 | Day 85
  Antibody titers at Day 85
RSV A serum neutralizing antibody titers at Day 113 Groups 2 and 4 | Day 113
  Antibody titers at Day 113
RSV B serum neutralizing antibody titers at Day 113 Groups 2 and 4 | Day 113
  Antibody titers at Day 113

SECONDARY OUTCOMES:
Anti- hepatitis B surface antigen (HBsAg) Immunoglobulin g (IgG) antibody (A)b concentrations ≥ 10 milli international units per milliliter (mIU/mL) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti- polyribosylribitol phosphate (PRP) Ab concentrations ≥ 0.15 micrograms per milliliter (µg/mL) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti-poliovirus types (1, 2, and 3) Ab titers ≥ 1:8 Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti-pertussis Ab concentrations pertussis toxin, filamentous hemagglutinin , pertactin, fimbriae (PT, FHA, PRN, FIM) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti-diphtheria Ab concentrations ≥ 0.1 IU/mL Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti-tetanus Ab concentrations ≥ 0.1 IU/mL Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti-pneumococcal Ab concentrations measured by electrochemiluminescence (ECL) for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F and 33F Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Anti-measles Ab concentrations ≥ 255 mIU/mL Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Anti-mumps Ab concentrations ≥ 10 antibody units (AbU/mL) Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Anti-rubella Ab concentrations ≥ 10 IU/mL Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Anti-varicella Ab concentrations ≥ 5 glycoprotein enzyme-linked immunosorbent assay (gpELISA) units/mL Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody 28 days after the 12 month routine vaccinations
Anti-pneumococcal Ab concentrations measured by ECL Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Descriptive: Anti-PRP Ab concentrations (µg/mL) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-diphtheria Ab concentrations (IU/mL) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-diphtheria Ab concentrations ≥ 0.01 IU/mL Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-tetanus Ab concentrations (IU/mL) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-tetanus Ab concentrations ≥ 0.01 IU/mL Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-HBsAg Ab concentrations (mIU/mL) Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-HBsAg Ab concentrations ≥ 100 mIU/mL Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-poliovirus types (1, 2, and 3) Ab titers Cohort 1 | 28 days after the 6 month routine vaccinations
  Antibody titers 28 days after the 6 month routine vaccinations
Descriptive: Anti-measles Ab concentrations (mIU/mL) Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Descriptive: Anti-mumps Ab concentrations (AbU/mL) Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Descriptive: Anti-rubella Ab concentrations (IU/mL) Cohort 2 | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
Descriptive: Anti-varicella Ab concentrations (gpELISA units/mL) | 28 days after the 12 month routine vaccinations
  Antibody titers 28 days after the 12 month routine vaccinations
RSV A serum neutralizing antibody titers by baseline serostatus at Day 1 Cohort 1 and Cohort 2 | Day 1
  Antibody titers at Day 1
RSV B serum neutralizing antibody titers by baseline serostatus at Day 1 Cohort 1 and Cohort 2 | Day 1
  Antibody titers at Day 1
RSV A serum neutralizing antibody titers by baseline serostatus 28 days post-dose 2 1 Cohort 1 and Cohort 2 | 28 days post-dose 2
  Antibody titers 28 days post-dose 2
RSV B serum neutralizing antibody titers by baseline serostatus 28 days post-dose 2 Cohort 1 and Cohort 2 | 28 days post-dose 2
  Antibody titers 28 days post-dose 2
Presence of solicited administration site reactions within 21 days after each investigational medicinal product (IMP) administration Cohort 1 and Cohort 2 | 21 days after each IMP administration
  Number of participants experiencing solicited administration site reactions
Presence of solicited systemic reactions within 21 days after each IMP administration Cohort 1 and Cohort 2 | 21 days after each IMP administration
  Number of participants experiencing solicited systemic site reactions
Presence of unsolicited systemic adverse events (AEs) reported in the 30 minutes after each study intervention administration Cohort 1 and Cohort 2 | Within 30 minutes after each study intervention administration
  Number of participants experiencing unsolicited systemic adverse events
Presence of unsolicited AEs within 28 days after each study intervention administration Cohort 1 and Cohort 2 | Within 28 days after each study intervention administration
  Number of participants experiencing unsolicited AEs
Presence of medically attended adverse events (MAAEs) throughout the study Cohort 1 and Cohort 2 | Throughout the study, approximately 9 months
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) throughout the study Cohort 1 and Cohort 2 | Throughout the study, approximately 9 months
  Number of participants experiencing SAEs
Presence of adverse events of special interest (AESIs) throughout the study Cohort 1 and Cohort 2 | Throughout the study, approximately 9 months
  Number of participants experiencing AESIs

CONTACTS AND LOCATIONS:
Locations (72):
- United States (66):
  - Alabama Clinical Therapeutics - Birmingham - St. Vincent's Drive- Site Number : 8400007, Birmingham, Alabama
  - South Alabama Medical Clinic- Site Number : 8400065, Grand Bay, Alabama
  - MedPharmics - Mobile - Dauphin Street- Site Number : 8400017, Mobile, Alabama
  - Northwest Arkansas Pediatric Clinic- Site Number : 8400002, Fayetteville, Arkansas
  - Alliance Research Institute - Bell Gardens - Garfield Avenue- Site Number : 8400040, Bell Gardens, California
  - Matrix Clinical Research - Huntington Park- Site Number : 8400018, Huntington Park, California
  - Paradigm Clinical Research Centers- Site Number : 8400059, La Mesa, California
  - Matrix Clinical Research - Los Angeles- Site Number : 8400008, Los Angeles, California
  - Kaiser Permanente - Oakland Medical Center- Site Number : 8400047, Oakland, California
  - Stanford University Medical Center CTRU - 800 Welch Road- Site Number : 8400070, Palo Alto, California
  - Kaiser Permanente - Sierra Gardens- Site Number : 8400063, Roseville, California
  - Kaiser Permanente - Point West Medical Offices- Site Number : 8400064, Sacramento, California
  - Kaiser Permanente - San Jose Medical Center- Site Number : 8400060, San Jose, California
  - Kaiser Permanente - Santa Clara Medical Center- Site Number : 8400061, Santa Clara, California
  - Integrated Clinical Research LLC- Site Number : 8400036, Sherman Oaks, California
  - Kaiser Permanente - Walnut Creek Medical Center- Site Number : 8400062, Walnut Creek, California
  - Velocity Clinical Research - Washington DC- Site Number : 8400050, Washington D.C., District of Columbia
  - Prohealth Research Center- Site Number : 8400068, Doral, Florida
  - The Medici Medical Research- Site Number : 8400055, Hollywood, Florida
  - Dade Research Center- Site Number : 8400014, Miami, Florida
  - Riveldi Biomedical Research and Associates - Miami Lakes- Site Number : 8400015, Miami Lakes, Florida
  - SEC Clinical Research - Pensacola- Site Number : 8400034, Pensacola, Florida
  - PAS Research- Site Number : 8400005, Tampa, Florida
  - Leavitt Women's Healthcare- Site Number : 8400009, Idaho Falls, Idaho
  - Velocity Clinical Research - Sioux City- Site Number : 8400054, Sioux City, Iowa
  - Alliance for Multispeciality Research - El Dorado- Site Number : 8400019, El Dorado, Kansas
  - University of Kentucky Chandler Medical Center- Site Number : 8400051, Lexington, Kentucky
  - Velocity Clinical Research - New Orleans- Site Number : 8400058, New Orleans, Louisiana
  - Research Works INC- Site Number : 8400044, New Orleans, Louisiana
  - Velocity Clinical Research - Gulfport- Site Number : 8400011, Gulfport, Mississippi
  - QPS Bio-Kinetic Clinical Applications- Site Number : 8400046, Springfield, Missouri
  - Boeson Research - Great Falls- Site Number : 8400041, Great Falls, Montana
  - Boeson Research - Missoula- Site Number : 8400006, Missoula, Montana
  - Velocity Clinical Research - Grand Island- Site Number : 8400016, Grand Island, Nebraska
  - Midwest Childrens Health Research Institute- Site Number : 8400038, Lincoln, Nebraska
  - Velocity Clinical Research - Omaha- Site Number : 8400001, Omaha, Nebraska
  - PAS Research - Henderson- Site Number : 8400049, Henderson, Nevada
  - NYU Langone Cardiothoracic Surgery Associates - Garden City- Site Number : 8400048, Garden City, New York
  - Summerwood Pediatrics- Site Number : 8400021, Liverpool, New York
  - SUNY Upstate Medical University - Syracuse- Site Number : 8400029, Syracuse, New York
  - Dayton Clinical Research- Site Number : 8400030, Dayton, Ohio
  - Ohio Pediatrics - Dayton- Site Number : 8400033, Dayton, Ohio
  - Senders Pediatrics- Site Number : 8400022, South Euclid, Ohio
  - Cyn3rgy Research- Site Number : 8400053, Gresham, Oregon
  - Square-1 Clinical Research- Site Number : 8400031, Erie, Pennsylvania
  - Pas Research - Pittsburgh- Site Number : 8400043, Pittsburgh, Pennsylvania
  - Neighbors Pediatrics- Site Number : 8400072, Charleston, South Carolina
  - Tribe Clinical Research - Greenville - Verdae Boulevard- Site Number : 8400012, Greenville, South Carolina
  - South Texas Clinical Research- Site Number : 8400004, Corpus Christi, Texas
  - Javara - Privia Medical Group North Texas - Dallas- Site Number : 8400003, Dallas, Texas
  - PAS Research - Children's Care Clinic- Site Number : 8400035, Edinburg, Texas
  - Helios Clinical Research - Fort Worth - 8th Avenue- Site Number : 8400020, Fort Worth, Texas
  - Ventavia Research Group - Houston - North Loop West- Site Number : 8400010, Houston, Texas
  - The University of Texas Health Science Center- Site Number : 8400037, Houston, Texas
  - DM Clinical Research - Houston - Jones Road- Site Number : 8400052, Houston, Texas
  - Mercury Clinical Research - Houston - Savoy Drive- Site Number : 8400045, Houston, Texas
  - La Providence Pediatrics & Family Clinics- Site Number : 8400039, Houston, Texas
  - Houston Clinical Research Associates- Site Number : 8400013, Houston, Texas
  - University of Texas Medical Branch at Galveston- Site Number : 8400057, League City, Texas
  - Maximos Ob/Gyn- Site Number : 8400024, League City, Texas
  - Research Your Health- Site Number : 8400066, Plano, Texas
  - Pediatric Center - Richmond- Site Number : 8400032, Richmond, Texas
  - North Houston Internal Medicine & Pediatric Clinic- Site Number : 8400025, Tomball, Texas
  - Utah Valley Pediatrics - Orem- Site Number : 8400067, Orem, Utah
  - Ogden Clinic - Mountain View - CCT Research- Site Number : 8400056, Pleasant View, Utah
  - Wee Care Pediatrics - Roy- Site Number : 8400071, Roy, Utah
- Mexico (3):
  - Investigational Site Number : 4840001, Mexico City, Mexico City
  - Investigational Site Number : 4840002, Temixco, Morelos
  - Investigational Site Number : 4840004, Mexico City
- Puerto Rico (3):
  - Investigational Site Number : 6300001, Caguas
  - Investigational Site Number : 6300003, Ponce
  - Investigational Site Number : 6300004, Trujillo Alto

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAD00016 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25734&tenant=MT_SNY_9011